CLINICAL TRIAL: NCT05479552
Title: A Diagnostic Test for Dementia With Lewy Bodies
Status: Active, not recruiting | Type: Observational
Sponsor: CND Life Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 101; R44AG076072 (NIH)
Record Dates: First submitted 2022-07-22; First posted 2022-07-29 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: MCI-AD, Early Stage Alzheimer's Disease; MCI-DLB, Early Stage Dementia With Lewy Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCI-AD: Will be diagnosed using 'preclinical AD' criteria of mild cognitive impairment supported by a positive biomarker for AD. MCI defined as: 1. History of cognitive decline, noticed by either the patient, family member(s) or a medical practitioner but still independent in most complex daily activities. 2. Documentation of cognition not normal e.g., by MoCA or neuropsychological testing; 3. Does not meet the definition of dementia with MOCA <18 or global CDR 1 or greater (although exceptions may exist with appropriate justification). 4. Supportive AD biomarker (has positive biomarkers for both Aβ and neuronal injury using CSF or neuroimaging).
  Interventions: Diagnostic Test: Syn-One Test
- MCI-DLB: Will be diagnosed as prodromal probable MCI-DLB based on consensus criteria using 2 or more core clinical features of DLB (with or without the presence of biomarkers) or 1 or more core clinical features with 1 or more indicative biomarkers (reduced dopamine transporter uptake in basal ganglia demonstrated by SPECT or PET reduced Iodine-MIBG uptake on myocardial scintigraphy, PSG confirmation of REM without atonia).
  Interventions: Diagnostic Test: Syn-One Test

INTERVENTIONS:
Diagnostic Test: Syn-One Test — CND Life Sciences is expanding the utility of its diagnostic technology, the Syn-One Test, to pathologically distinguish between early DLB and Alzheimer's disease to prevent misdiagnoses and establish the relationship between progression and α-synuclein deposition by measuring α- synuclein accumulation in patient's nerve fibers using a simple skin punch biopsy.

SUMMARY:
The Syn-D Study will be evaluating α-synuclein in patients with suspected MCI-AD and MCI-DLB. Using a simple diagnostic test will improve clinical accuracy in diagnosing, earlier diagnosis, and distinguish between neurodegenerative diseases.

DETAILED DESCRIPTION:
In collaboration with approximately 10 centers that specialize in DLB and dementia we will recruit a total of 80 individuals for the study: 40 subjects with suspected MCI-DLB and 40 with suspected MCI-AD will be recruited. All subjects will be enrolled into a 12 month longitudinal study where skin biopsies will be performed at 3 sites on each patients at 12 month intervals (baseline and 1 year). Detailed quantified examination, cognitive evaluation, history, and questionnaires will be performed at each visit and will be reviewed by a central panel of disease experts to confirm the diagnosis.

Subjects enrolled in the study will have baseline evaluations and follow up visits at 12 months to define any changes to clinical diagnosis. Skin biopsies will be repeated at the 12 month follow up visit to determine the rate of P-SYN accumulation over time and rates of nerve fiber degeneration within punch skin biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 50 to 85 years of age
2. Clinical diagnosis of mild cognitive impairment, and a presumed etiology of DLB or AD at enrollment

Exclusion Criteria:

1. Clinical evidence of severe peripheral vascular disease (Fazekas score of ≥ 3, or a large vessel stroke of ≥ 2 cm, history of ulceration, poor wound healing, vascular claudication)
2. Clinically active coronary artery or cerebrovascular disease
3. Current smoker or alcoholism
4. History of allergic reaction to local anesthesia (for biopsy collection)
5. Use of anticoagulants (aspirin or Plavix alone is allowed)
6. Significantly impaired wound healing or history of scarring or keloid formation

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex is determined by gender at birth.
Study Population: The subjects evaluated in the protocol will have a diagnosis of mild dementia with Lewy bodies (MCI-DLB) or mild Alzheimer's disease (MCI-AD). Patients will be evaluated at Baseline and 12 months. A total of 80 individuals will be enrolled, 40 with MCI-DLB and 40 with MCD-AD, with roughly equal representation of men and women.
  All subjects will undergo screening evaluation that includes a thorough medical history, physical and neurologic examination and review of available medical records, laboratory studies, neuroimaging and sleep laboratory studies.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
This is a prospective longitudinal study of individuals with neurodegenerative DLB and AD disorders to improve the diagnostic precision and utility of the Syn-One TestTM. | 2 years
  To pathologically distinguish DLB from AD early in the course of the disease using the Syn-One TestTM, confirming disease diagnosis through prospective clinical assessments and follow up biopsy analyses over 12 months.
This is a prospective longitudinal study of individuals with neurodegenerative DLB and AD disorders to improve the diagnostic precision and utility of the Syn-One TestTM. | 2 years
  To define the rates of neuronal degeneration in DLB through systematic pathological quantitation of skin biopsies measuring P-SYN deposition and cutaneous nerve fiber degeneration, compared to AD, and correlating pathological findings with clinical assessments over the course of 12 months.

SECONDARY OUTCOMES:
Secondary Aim 1 | 2 years
  The outcome measure will be an ordinal quantitation of P-SYN deposition within skin biopsies. The primary endpoint for is sensitivity and specificity of results in DLB and AD. We predict that a threshold of P-SYN >0 is a "positive" result and will separate DLB from AD using dichotomous measures, but ROC curve analysis will be performed to maximize sensitivity and specificity using continuous quantitative measurement of P- SYN.
Secondary Aim 2 | 2 years
  Will include P-SYN deposition, SGNFD, PMNFD and IENFD as continuous variables for statistical analysis. Data will be compared first using repeated measures Analysis of Covariance (ANCOVA), with DLB as the predictor variable. The primary dependent variable is the quantitative measure of P-SYN deposition.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Levine, MD, Principal Investigator — CND Life Sciences
Locations (12):
- United States (12):
  - CND Life Sciences, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - CenExel RMCR, Englewood, Colorado
  - University of Miami, Boca Raton, Florida
  - Neurology One, Winter Park, Florida
  - Ochsner Research, New Orleans, Louisiana
  - Mass General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Headlands Research, Plymouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with researchers that are involved in the study.

REFERENCES:
- [Background] Gibbons CH, Freeman R, Bellaire B, Adler CH, Moore D, Levine T. Synuclein-One study: skin biopsy detection of phosphorylated alpha-synuclein for diagnosis of synucleinopathies. Biomark Med. 2022 May;16(7):499-509. doi: 10.2217/bmm-2021-0646. Epub 2022 Mar 11. PMID 35272481
- [Derived] Gibbons CH, Galasko D, Press D, Claassen D, Levine T, Freeman R. The Syn-D study: detection of cutaneous phosphorylated alpha-synuclein in mild cognitive impairment a trial protocol. Biomark Med. 2025 Jul;19(13):501-508. doi: 10.1080/17520363.2025.2520154. Epub 2025 Jun 16. PMID 40523872